CLINICAL TRIAL: NCT00003200
Title: Taxotere Plus Concurrent Radiotherapy After Induction Chemotherapy for Squamous Cell Carcinoma of the Head and Neck (TAXT-XRT)
Brief Title: Chemotherapy Plus Radiation Therapy in Treating Patients With Squamous Cell Cancer of the Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert I. Haddad, MD, Haddad, Robert MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 95-041; P30CA006516 (NIH); NCI-G98-1382
Record Dates: First submitted 1999-11-01; First posted 2004-08-13 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Docetaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Taxotere (Experimental): After the screening procedures confirm participation in the research study:
  * Taxotere-Administered weekly for 1 hour (6 doses)
  * Radiation Therapy (XRT) -5 days a week for 6 weeks
  * Exam under anesthesia
  * Neck Dissection (if indicated)
  Interventions: Drug: Taxotere; Radiation: Radiation therapy

INTERVENTIONS:
Drug: Taxotere
  Other Names: Docetaxel
Radiation: Radiation therapy

SUMMARY:
The purpose of this research study is to develop a new chemo radiotherapy regimen for the treatment of cancer of the head and neck for patients who have received induction chemotherapy; and to determine the highest dose of Taxotere which can be safely given together with radiotherapy.

DETAILED DESCRIPTION:
In this investigational research study investigators are attempting to develop a new chemo radiotherapy regimen in which radiotherapy and Taxotere will be combined after having received induction chemotherapy. Taxotere has never been given together with radiotherapy, the highest dose of Taxotere that can be safely used in this setting in unknown. Taxotere will be added to radiotherapy gradually as each subsequent group of 3-5 patients gets a larger dose. Taxotere doses will be increased until certain toxicities occur. This will help investigators determine the best way to combine Taxotere with radiotherapy and to use that knowledge to treat other patients with tumors like yours.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathology: Histologic documentation of squamous cell carcinoma of the head and neck or its variants (lymphoepithelioma, undifferentiated epidermoid carcinoma, etc)
* Stage: Patients can be entered on this protocol after initial induction therapy, if prior to the induction regimen, they were previously untreated Stage III or IV (MO) SCCHN. This excludes patients with exophytic T3N0 tumors or T1N1 lesions at the onset of induction therapy. Evaluable disease during induction therapy is required.

  --Required Prior therapy: Patients entered on this protocol must have received therapy with one of the following induction regimens, except as modified for toxicity:
  * PF: Cisplatin ≥ 80 mg/M2?course and FUra ≥ 1000 mg/M2/day for ≥ 4 days every ≤ 4 week
  * CF: Carboplatinum ≥ 300 mg/M2/course and FUra ≥1000mg/M2/day for ≥4 days for ≤ 4 week
  * PFL5: Cisplatin ≥ 25 mg/M2/day over 5 days, FUra ≥ 800mg/M2/day days 2-5 (4 days) and Leucovorin ≥ 500 mg/M2/day over 5 days, every 4 weeks.
  * TPF: Taxotere, Cisplatin ≥ 100 mg/M2/day over 5 days, FUra ≥ 700 mg/M2?day days 2-5 (4 days)
  * Patients treated as above are eligible provided that they receive no more than three cycles or, if not responding after 2 cycles; or 1 cycle with progressive disease p. 35 of archive doc
* Other Malignancies:

  * Patients with previous head and neck cancer are ineligible, except patients who were treated with surgery as the sole modality 2 years prior to study entry.
  * Patients with concurrent malignancy of any site, except limited basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix are ineligible.
  * Patient with any non-SCCHN malignancy within 5 years of study entry, except curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix are ineligible.
* Other Prior Therapy: Patients who were previously treated with radiotherapy for SCCHN are not eligible. Patients treated with any form of prior chemotherapy , other than induction therapy described in section 3.21 within the last 5 years are not eligible. Hormonally treated patients are eligible.
* Performance: Patients must meet the following performance criteria:

  * Performance status: 2 ECOG. Complete recovery from previous diagnostic or therapeutic procedures is required.
  * Nutritional status: Adequate and nutritionally balances enteral intake (1,800 kcal/day). Patients requiring intravenous alimentation as primary source of calories are excluded from this study. Patients who experiences a weight loss of more than 20% of their body weight in the three months preceding presentation are ineligible. Patients with persistent diarrhea are ineligible.
  * Life Expectancy: Longer than 3 Months
  * Women of child bearing potential must not be pregnant by history or lactating at the time of entry on this protocol and men and women of child bearing potential must be requested to use an accepted and effective method of birth control during therapy.
* Organ Function: Biochemical and hematological parameters (obtained within 2 weeks of study entry) as follows:

  * Hepatic: SGOT < 1.5 x ULN and Alkaline Phosphatase < 2.5x ULN for entry. Total Bilirubin and SGOT must be ≤ 2 x ULN as an isolated value. Alkaline phosphatase must be ≤ 2.5 x ULN as an isolated value.
  * Hematologic: WBC 4,000/mm3 or a normal absolute neutrophil count (ANC); Platelet count 100,000/mm3, Hemoglobin 10 gm/dl (transfusion to bring the hemoglobin to or above this level is permitted if clinically indicated, however, transfusions should not be used solely in order to eligibility criteria)
  * Neurologic: Peripheral neuropathy of any etiology must not exceed grade 1.
  * Cardiovascular/Pulmonary: No acute cardiac dysrhythmias or unstable cardiac condition such as angina
  * Other: Lack of other serious illness or medical condition
* Allergies: Patients with prior allergy to polysorbate 80 (see appendix) are ineligible
* Informed Consent: Patients must give written informed consent
* Follow-up: All patients must be available for monthly evaluation and restaging by the head and neck cancer clinic on therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 1995-10; Primary Completion 2006-10 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
MTD of weekly Taxotere | 6 Weeks
Number of Participants of with Severe Adverse Events | 6 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marshall R. Posner, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Harvard Community Health Plan, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No